CLINICAL TRIAL: NCT05942196
Title: Validation du Questionnaire d'Evaluation de la Perception de l'Activité Physique (EPAP) adapté à la Lombalgie Chronique
Brief Title: Validation of the Evaluation of the Perception of Physical Activity Questionnaire Adapted to Chronic Low Back Pain
Acronym: EPAP-LOMB
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Centre de Rééducation Fonctionnelle de Notre-Dame, Chamalières (Unknown)
Responsible Party: Sponsor
Other Study IDs: RNI 2023 COUDEYRE; 2023-A00504-41 (Other: ANSM)
Record Dates: First submitted 2023-06-14; First posted 2023-07-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2024-07

CONDITIONS: Chronic Low Back Pain
Keywords: Chronic low back pain; Physical activity; Patient-reported outcome; Facilitators; Barriers; Psychometric properties
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Physical exercise has a fundamental position in the chronic low back pain treatment. However, the physical activity level is often low in these patients and the adherence to the care program is not enough in the long term. The French Evaluation of the Perception of Physical Activity (EPPA) is a valid and reliable questionnaire, developed by N. Coste et al in 2020, that assesses the perceived barriers to and facilitators of physical activity in patients with knee osteoarthritis. To our knowledge, there is no valid and reliable instrument allowing such an assessment in chronic low back pain.

The main objective of this study is to adapt the EPPA to chronic low back pain and to evaluate its psychometric properties.

This validation would allow its use in current practice to adapt the care strategy, to personalize rehabilitation of each patient with chronic low back pain in order to have a better adherence to rehabilitation programs.

DETAILED DESCRIPTION:
The EPPA was adapted to chronic low back pain and named EPPA-LOMB. It comprises 26 items.

Patients with chronic low back pain will be recruited during a medical consultation in the Physical Medicine and Rehabilitation Department of the University Hospital of Clermont-Ferrand and the Notre-Dame Functional Rehabilitation Center of Chamalières (France); or the first day of a functional spine rehabilitation program (3-week program in a day hospital) in the Physical Medicine and Rehabilitation Department of the University Hospital of Clermont-Ferrand.

Patients will be asked to complete a series of questionnaires after completing the non-opposition form. The management of non-specific chronic low back pain also requires evaluation through questionnaires, in accordance with the usual practices of the services participating in the study. No intervention will be taken.

All patients will complete questionnaires at inclusion.

Patients included during a medical consultation will receive an e-mail to complete online the EPPA-LOMB and visual analogic scales on pain and level of physical activity, 7 days after inclusion.

Patients included the first day of a functional spine rehabilitation program will complete questionnaires at the end of the program, 21 days after inclusion. They will be seen 3 months after their discharge during a follow-up medical consultation and will complete another time the questionnaires. Only patients not included in the study E-lombactifs (NCT04264949) will complete the questionnaire at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years old and older)
* Patients with chronic low back pain evolving for at least 3 months, with a diagnosis confirmed by the French Health Authority and the classification from the French and European recommendations, that is lumbar pain, without red flags, with a possible pain radiculopathy
* Acceptance to participate in the study.
* Capable of providing informed consent to participate in this study.

Exclusion Criteria:

* Patients not diagnosed according to the French Health Authority and the classification from the French and European recommendations
* Refusal to participate
* Patients in the incapacity to answer the questionnaires
* Patients with a medical contraindication to physical activity
* Patients under guardianship, or protection of justice.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic low back pain seen in the Physical Medicine and Rehabilitation Department of the University Hospital of Clermont-Ferrand and in the Notre-Dame Functional Rehabilitation Center of Chamalières (France).
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
EPPA-LOMB | 0 day
  Acceptability, internal validity, convergent validity, validity of structure against external criteria of the French questionnaire EPPA-LOMB.
Change of EPPA-LOMB from baseline at 7 days | 0 day, 7 days
  Test-retest reliability of the French questionnaire EPPA-LOMB.
Change of EPPA-LOMB from baseline at 21 days | 0 day, 21 days
  Responsiveness of the French questionnaire EPPA-LOMB.
Change of EPPA-LOMB from baseline at 3 months | 0 day, 3 months
  Responsiveness of the French questionnaire EPPA-LOMB.

SECONDARY OUTCOMES:
Visual analogic scale for physical activity | 0 day, 7 days, 21 days, 3 months
  Visual analogic scale for physical activity (VAS physical activity) from 0- no physical activity to 10-very intense physical activity
Visual analogic scale for pain | 0 day, 7 days, 21 days, 3 months
  Visual analogic scale for pain (VAS pain) from 0-no pain to 10-the worst pain
OSWESTRY Disability Index (ODI) | 0 day, 21 days, 3 months
  The functional disability is measured by the OSWESTRY Disability Index (ODI). Ten items rated from 0 to 5 compose a valid and reliable scale with a total score ranging between 0 and 50.
Fear Avoidance Belief Questionnaire (FABQ) | 0 day, 21 days, 3 months
  The fears and the faiths are measured by the Fear Avoidance Belief Questionnaire (FABQ). The FABQ can help predict those that have a high pain avoidance behavior. Clinically, these people may need to be supervised more than those that confront their pain. The FABQ contains 2 scales: a work scale (FABQ-W) composed of 7 items and a physical activity scale (FABQ-PA) composed of 4 items. The two scales are scored separately. Higher FABQ scores indicate elevated fear-avoidance beliefs. "FABQ-W" has a point score that ranges from 0-42 points and "FABQ-PA" can range from 0-24 points.
Exercise Adherence Rating Scale (EARS) | 0 day, 21 days, 3 months
  The Exercise Adherence Rating Scale (EARS) is a reliable and validated psychometric assessment questionnaire that assesses adherence to prescribed physical exercise in chronic low back pain.A 6-item adherence scale assess adherence to prescribed home exercise. These six items are scored on a 5-point Likert scale (0 = completely agree, 4 = completely disagree). Items 2, 3 and 5 are negatively worded questions. Therefore, higher sum scores (0-24) indicate greater exercise adherence by reversing scores of Items 1, 4, and 6. Ten supplementary items assess reasons for adherence and non-adherence.
the Hospital Anxiety and Depression Scale (HADS) | 0 day, 21 days, 3 months
  The knowledge of emotional state is measured by the Hospital Anxiety and Depression Scale (HADS). The HADS is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. HADS gives clinically meaningful results as a psychological screening tool and can assess the symptom severity and caseness of anxiety disorders and depression in patients with illness and the general population. The questionnaire, comprising fourteen items. Each item is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.
Socio-demographic and medical characteristics. | 0 day
  Gender, age, body mass index, time since first symptoms, family situation, edicational level, type and frequency of regular physical activities, type and frequency of regular leisure activities, type of treatment provided for chronic low back pain, comorbidity, antalgic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Emmnauel COUDEYRE, Principal Investigator — ecoudeyre@chu-clermontferrand.fr
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Oliveira CB, Maher CG, Pinto RZ, Traeger AC, Lin CC, Chenot JF, van Tulder M, Koes BW. Clinical practice guidelines for the management of non-specific low back pain in primary care: an updated overview. Eur Spine J. 2018 Nov;27(11):2791-2803. doi: 10.1007/s00586-018-5673-2. Epub 2018 Jul 3. PMID 29971708
- [Background] Bailly F, Trouvin AP, Bercier S, Dadoun S, Deneuville JP, Faguer R, Fassier JB, Koleck M, Lassalle L, Le Vraux T, Liesse B, Petitprez K, Ramond-Roquin A, Renard JF, Roren A, et al. Recommandations et arbre décisionnel sur la prise en charge de la lombalgie avec ou sans radiculalgie. Revue du Rhumatisme. 2022 ; 89 : 345-353.
- See also: French recommendations for chronic low back pain — https://pubmed.ncbi.nlm.nih.gov/38693474/
- See also: French Health Authority recommendations for the diagnosis of chronic low back pain — https://www.has-sante.fr/jcms/c_2961499/fr/prise-en-charge-du-patient-presentant-une-lombalgie-commune